CLINICAL TRIAL: NCT00283270
Title: A Randomised Controlled Trial on the Effectiveness of Screening and Brief Counselling for Elderly Patients With Psychological Problems in Primary Care.
Brief Title: Effectiveness of Screening and Counselling for Elderly With Psychological Problems
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Health Care and promotion Fund, the Governement of the Hong Kong SAR. (Unknown)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RESCEP; HCPF 218016
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Last update posted 2006-01-27 (Estimated); Status verified 2005-12

CONDITIONS: Mental Illness
Keywords: Mental health; Screening; Elderly; Chinese; Problem-solving counselling
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being

INTERVENTIONS:
Behavioral: Brief counselling
Behavioral: Behavior

SUMMARY:
The aim of the study is to test whether screening followed by brief problem-solving counselling in primary care could improve the quality of life of elderly patients with undiagnosed psychological problems. We hypothesize that undiagnosed psychological problems detectable by screening are common in the elderly and brief counselling could improve the quality of life of these patients.

DETAILED DESCRIPTION:
Objectives: The aim of the study is to test if screening followed by brief problem-solving counselling by primary care doctors can improve the health-related quality of life (HRQOL) of elderly patients with previously undiagnosed psychological problems. It will also find out the effects of undiagnosed psychological problems on HRQOL and consultation rates of elderly patients.

Design, Setting & Subjects: This is a prospective single-blinded randomised controlled trial on 450 patients aged 60 or above attending a Government General Outpatient Clinic in Hong Kong, who have been screened for psychological problems.

Methods: Elderly patients attending the General Outpatient Department of the Ap Lei Chau Clinic who are not known to have the diagnosis of psychological problems with the Hospital Anxiety & Depression Scale (HADS) were screened in order to recruit 300 subjects who are screened positive for undiagnosed psychological problems will be randomised into the counselling or no-counselling groups, and 150 subjects who are screened negative for psychological problems will be selected as normal controls

Interventions: The counselling group will receive brief problem-solving counselling from a trained primary care doctor in addition to their usual medical care; the no-counselling group will receive general health education and their usual medical care; and the normal control group will continue with their usual care only.

Main Outcome Measures: Health-related quality of life measured by the SF-36, the HADS scores and consultation rates. The baseline and changes in outcomes of the three groups will be compared at 0, 6, 12, 36 and 52 weeks after screening.

Conclusions: The results will provide evidence on whether screening followed by brief problem-solving counselling in primary care is effective in improving quality of life and reducing consultation rates for the elderly with undiagnosed psychological problems.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 60 or above
2. Attending the study primary care clinic
3. No known diagnosis of psychological problem
4. Written consent provided

Exclusion Criteria:

1. Known psychological disease diagnosed by a registered practitioner
2. Taking any psychotropic drug prescribed by a registered practitioner of Western medicine within the last year;
3. Has suicidal plan or strong suicidal thought;
4. Has psychotic symptom;
5. any impairment in cognitive function; or
6. any communication problem
7. refuses to participate

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450
Dates: Start 2002-11; Study Completion 2005-08

PRIMARY OUTCOMES:
Health-related quality of life scores
Hospital Anxiety and Depresssion scores

SECONDARY OUTCOMES:
Consultation rates

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L Lam, MD, Principal Investigator — The University of Hong Kong